CLINICAL TRIAL: NCT07102745
Title: HomeLink2: Reducing Posthospitalization Mortality Through Structured Home Care and Nutritional Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00449828; R01MH138270 (NIH)
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: HIV care post-hospitalization; Home-based care for HIV; Nutritional support for HIV; People living with HIV
MeSH Terms: interventions — Nutritional Support

STUDY DESIGN:
Intervention Model Description: Individually randomized, three arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (No Intervention): Participants in the standard of care arm will receive discharge care as routinely provided at Tshepong Hospital. This includes scheduling follow-up, which is usually two weeks following discharge and usually at the appropriate specialty clinic located at Tshepong Hospital.
- Home Visit Study Arm (Experimental): In addition to receiving the routine discharge care provided at Tshepong Hospital (as in the standard of care arm), participants in the home visit intervention arm will receive regular home visits every two weeks, starting one week after hospital discharge, for a total of 4 to 6 visits. Each visit will be conducted by a trained nurse-clinician and counselor, with the aim of building trust through continuity of care. During each visit, the team will provide clinical assessments, monitor vital signs, review medications with a focus on HIV treatment adherence, collect lab specimens if needed, and assess the home environment for safety and support. Psychosocial support will also be provided, including counseling on mental health, alcohol use, social support, and HIV-related challenges, using motivational interviewing techniques. Referrals will be made as needed for medical, mental health, or social services.
  Interventions: Behavioral: HomeLink
- Home Visit Plus Nutritional Support Arm (Experimental): Home visits will be conducted for the 'home visit study arm.' In addition, participants randomized to the home visit plus nutritional support study arm will receive food parcels. Food parcels will be provided by the Perinatal HIV Research Unit (PHRU) study team in 3 standardized and pre-packaged deliveries at weeks 1, 5, and 9.
  Interventions: Behavioral: HomeLink; Behavioral: HomeLink Plus Nutritional Support

INTERVENTIONS:
Behavioral: HomeLink — HomeLink is a structured post-discharge home-based care program for people living with HIV, designed to improve health outcomes after hospital discharge. Starting one week after discharge, trained nurse-clinician and counselor teams conduct regular home visits every two weeks for up to six visits. During these visits, the team will provide clinical assessments, medication adherence support, psychosocial counseling, specimen collection, and home safety evaluations. The intervention aims to offer personalized, continuous care that addresses medical, psychological, and social needs in the participant's home environment, enhancing recovery and reducing post-hospital mortality.
  Arms: Home Visit Plus Nutritional Support Arm; Home Visit Study Arm
Behavioral: HomeLink Plus Nutritional Support — This intervention combines the HomeLink home-based care program with the provision of nutritional support through food parcels. Participants receive food parcels designed to address nutritional needs and support overall health and recovery. The combined approach aims to improve post-discharge outcomes by addressing both medical and nutritional factors contributing to patient well-being.
  Arms: Home Visit Plus Nutritional Support Arm

SUMMARY:
People living with HIV (PLWH) are at high risk of poor health outcomes after being discharged from the hospital. This study is designed to test whether providing structured care at home-either with or without nutritional support-can help reduce the risk of death within six months of discharge and improve long-term health outcomes.

The investigators are conducting a randomized clinical trial to evaluate the effectiveness of home-based care on post-hospital recovery. Participants are randomly assigned to one of three groups: (1) standard post-discharge care, (2) home-based care that includes medical assessments, support for taking HIV medications (adherence support), and psychosocial counseling, or (3) the same home-based care plus food parcels to support nutrition.

This is a three-arm, individually randomized clinical trial and a type-1 hybrid implementation-effectiveness study, which means the investigators are not only testing whether the interventions improve health outcomes, but also examining how the interventions are delivered and whether the interventions are practical and acceptable in real-world settings. The trial begins with a pilot phase to test the investigators enrollment procedures and improve baseline data collection.

In addition to measuring whether the interventions reduce the risk of death, the study will assess how many people receive the intervention, whether it is acceptable to patients and families, and how consistently it is delivered. The investigators are also evaluating the economic impact of illness, hospitalization, and death on households, and analyzing the cost and resource needs of delivering home-based care, with or without food support.

The investigators goal is to provide evidence that can improve care for people living with HIV after hospital discharge. If effective, this approach may be applied more broadly to improve outcomes for other high-risk patients in similar settings. Findings from the study will be used to inform health policy and clinical practice, particularly in areas with limited resources and high HIV burden.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection (either diagnosed during or prior to hospital admission), consisting of any clinical documentation, including a chart note of HIV positivity, Ritonavir-boosted darunavir (RVD) positivity, or antiretroviral therapy (ART) regimen documentation/prescription
* ≥18 years old as per hospital file or government issued document
* Self-report that the participant resides within Matlosana sub-district
* Admitted to an adult internal medicine ward at Tshepong Hospital
* Have spent at least 2 nights in the hospital prior to recruitment to the trial.
* Agree to post-discharge follow-up, including home visits
* Are able to provide informed consent or if lacking capacity to provide consent at the time of recruitment, as determined by the study team, have a next of kin able to provide informed consent.

Exclusion Criteria:

* Admitted to a non-medical (i.e., surgical, psychiatric, etc.) ward, admitted for elective reasons, or admitted to facilitate onward transfer to another hospital
* Participant or next of kin unable to provide written informed consent in any of the languages of the informed consents or spoken by the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2028-09-04 (Estimated); Study Completion 2029-03-06 (Estimated)

PRIMARY OUTCOMES:
6-month all-cause mortality by intervention arm | 6 months post hospital discharge
  All-cause mortality at 6 months post-hospital discharge, comparing each intervention arm (HomeLink home visit, HomeLink plus nutritional support) separately and combined against standard discharge care.

SECONDARY OUTCOMES:
12-Month All-Cause Mortality | 12 months post hospital discharge
  Comparison of all-cause mortality at 12 months post-discharge between intervention arms and standard care.
Days of Rehospitalization | 12 months post hospital discharge
  Total number of days hospitalized during the 12-month follow-up period analyzed using negative binomial regression.
Time to First Care Visit | From discharge until first care visit within 12 months
  Time (measured in # of days) from hospital discharge to first care visit (home visit, fixed clinic, or fixed clinic only), analyzed using survival analysis methods.
Viral Load Suppression at 12 Weeks | 12 weeks post hospital discharge
  Proportion of participants with suppressed viral load at 12 weeks post-discharge by study arm.
Weight Change at 12 Weeks | From enrollment to 12 weeks post hospital discharge
  Comparison of weight change from enrollment to 12 weeks post-discharge between intervention arms. Weight will be measured in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Neil Martinson, Principal Investigator — Perinatal HIV Research Unit (PHRU); Christopher Hoffmann, Principal Investigator — Johns Hopkins University
Locations (1):
- Tshepong Hospital, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets including HIV status, viral load, clinical data, health service use, food security, social support, quality of life, participant health costs, HIV stigma, violence screening, health system trust, and weight measurements. Qualitative interview data will be stored securely and may be shared upon request under restricted access. Data will be date-offset to protect confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 6 to 24 months after completion of data collection, following cleaning, de-identification, and locking of datasets. Data will be stored and accessible for at least 10 years.
Access Criteria: Access will be granted to qualified researchers who submit a data use request to the Principal Investigator and obtain Institutional Review Board (IRB) approval for secondary analyses. Data access will be controlled through a repository (Dryad) that applies an independent review panel. Researchers will access de-identified and date-offset data and associated supporting documents via the repository under controlled conditions designed to protect participant privacy. Qualitative data will be accessed only by request and with restrictions.